CLINICAL TRIAL: NCT03106077
Title: Women's Triple-Negative First-Line Study: A Phase II Trial of Mirvetuximab Soravtansine in Patients With Localized Triple-Negative Breast Cancer (TNBC) With Tumors Predicted Insensitive to Standard Neoadjuvant Chemotherapy (NACT), Including a Lead-In Cohort to Establish Activity in Patients With Metastatic TNBC
Brief Title: Mirvetuximab Soravtansine as First Line in Treating Patients With Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0683; NCI-2018-01213 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0683 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Estrogen Receptor Negative; Folate Receptor Alpha Positive; HER2/Neu Negative; Progesterone Receptor Negative; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (mirvetuximab soravtansine) (Experimental): Patients receive mirvetuximab soravtansine IV over 2-3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Biological: Mirvetuximab Soravtansine
- Cohort B (mirvetuximab soravtansine) (Experimental): Patients receive mirvetuximab soravtansine IV over 2-3 hours on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unaccepted toxicity.
  Interventions: Biological: Mirvetuximab Soravtansine

INTERVENTIONS:
Biological: Mirvetuximab Soravtansine — Given IV
  Other Names: IMGN853; M9346A-sulfo-SPDB-DM4

SUMMARY:
This phase II trial studies how well mirvetuximab soravtansine works as first line in treating patients with triple negative breast cancer. Drugs used in chemotherapy, such as mirvetuximab soravtansine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* I. Determine if mirvetuximab soravtansine as a single agent is likely to induce response in at least 20% of patients with metastatic folate receptor (FR) alpha+ triple negative breast cancer (TNBC).
* II. Determine if mirvetuximab soravtansine as a single agent in the neoadjuvant setting will improve rates of excellent pathologic response (pathologic complete response [pCR]/residual cancer burden [RCB]-0 or RCB-I) from 5% to 20% in patients with high risk, chemotherapy insensitive, FRalpha+ TNBC.

SECONDARY OBJECTIVES:

* I. Determine the radiographic response rate as measured by ultrasound and/ or magnetic resonance imaging (MRI) (partial response + complete clinical response) for mirvetuximab soravtansine in chemotherapy insensitive, FRalpha

  + localized TNBC or using Response Evaluation Criteria in Solid Tumors (RECIST) criteria in patients with FRalpha+ advanced TNBC.
* II. Determine toxicity of 4 cycles of mirvetuximab soravtansine given in the neoadjuvant setting following anthracycline based therapy (Cohort B) and unrestricted cycles in patients receiving therapy in the advanced/metastatic setting (Cohort A).
* III. Determine disease free survival (DFS) at 3 years for patients treated with mirvetuximab soravtansine given in the neoadjuvant setting; progression free survival (PFS), duration of response (DOR) and overall survival at 3 years (overall survival [OS] at 3 years) in patients receiving therapy for advanced/ metastatic TNBC.
* IV. Compare disease response (as measured by pCR/RCB-I) in patients with FRalpha+ chemotherapy resistant disease treated on clinical trial with mirvetuximab soravtansine in the neoadjuvant setting to those with similar molecular features who receive standard taxane-based chemotherapy as the second phase of their NACT.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Confirmed invasive triple-negative breast cancer defined as estrogen receptor (ER) < 10%; progesterone receptor (PR) < 10% by immunohistochemistry (IHC) and HER2 0-1+ by IHC or 2+, fluorescence in situ hybridization (FISH) < 2, gene copy number < 4
* (For Cohort A) - Archived tissue available at pre-screening to confirm FR alpha+ breast cancer
* (For Cohort A) Archived tissue available pre-screening to confirm FR alpha+ breast cancer. (For Cohort B) Confirmed FRalpha+ breast cancer defined as low FRalpha expression: >= 25% of cells having >= 1+ expression
* (For Cohort A) Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST). (For cohort B) Clinical or radiologic primary tumor size of at least 1.5 cm prior to enrollment onto protocol 2014-0185 (ARTEMIS). Primary tumor of at least 1.0 cm or evidence of continued lymph node involvement by imaging (ultrasound or magnetic resonance imaging [MRI]) after adriamycin-based neoadjuvant therapy
* (For cohort B): Primary tumor sample collected before NACT started (on ARTEMIS) and underwent molecular testing for integral biomarkers including immunohistochemical assessment of FRalpha
* (For cohort A): No limit on prior therapies for metastatic disease. (Relapse of disease within 6 months of adjuvant or neoadjuvant chemotherapy is considered 1 line of therapy for metastatic disease). (For cohort B): received at least one dose of an anthracycline-based NACT. Patients are eligible if therapy was discontinued due to disease progression or therapy intolerance. Patients with disease progression on anthracycline-based therapy should be evaluated by the surgical team. If the patient is deemed inoperable at the time of evaluation, the patient may continue to undergo protocol therapy with a goal of reduction in tumor size to become operable. If the patient is deemed at high risk of becoming inoperable by the surgical team based upon tumor size or location, the patient will be considered ineligible for study and will be recommended to go to surgery
* (For cohort B): Primary tumor size of at least 1.0 cm by imaging (ultrasound or MRI) or evidence of continued lymph node involvement by imaging (ultrasound or MRI) after adriamycin-based neoadjuvant therapy
* (For cohort B): Baseline multigated acquisition (MUGA) or echocardiogram showing left ventricular ejection fraction (LVEF) >= 50% within 6 weeks prior to initiation of NACT
* (For both cohorts A and B): Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* (For both cohorts A and B): Platelets >= 100 x 10^9/L
* (For both cohorts A and B): Hemoglobin (Hb) > 9 G/dL
* (For both cohorts A and B): Total serum bilirubin =< 2.0 mg/dL
* (For both cohorts A and B): Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN) (=< 5 x ULN in patients with liver metastases)
* (For both cohorts A and B): International normalized ratio (INR) =< 2
* (For both cohorts A and B): Serum creatinine =< 1.5 x ULN
* (For both cohorts A and B): Serum albumin > 2
* Signed informed consent obtained prior to any screening procedures
* (For cohort A only): Time from prior therapy: a. Systemic anti-neoplastic therapy: five half-lives or four weeks, whichever is shorter. Hormonal therapy is not considered anti-neoplastic therapy. b. Radiotherapy: wide-field radiotherapy (e.g. > 30% of marrow-bearing bones) completed at least four weeks, or focal radiation completed at least two weeks, prior to starting study treatment
* (For cohort B only): Patients must have at least 3 and no more than 5 weeks between anthracycline-based therapy and start of treatment with mirvetuximab soravtansine
* (For both cohorts A and B): Patients must have resolution of toxic effect(s) of the most recent prior chemotherapy to grade 1 or less (except alopecia)
* (For both cohorts A and B): Women of child-hearing potential (WCBP) must have a negative pregnancy test within 3 days prior to the first dose of study treatment

Exclusion Criteria:

* Pregnant or lactating women
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* (For Cohort B only): Presence of metastatic disease or prior radiation therapy of the primary breast carcinoma or axillary lymph nodes
* Women of child-bearing potential (WCBP), defined as all women capable of becoming pregnant, won't use highly effective methods of contraception during the study and 12 weeks after. Highly effective contraception methods include combination of any two of the following:

  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Total abstinence or
  * Male/female sterilization
  * Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile, or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to study entry. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential
* Male patients whose sexual partner(s) are WCBP who are not willing to use adequate contraception, during the study and for 12 weeks after the end of treatment
* Patients with > grade 1 peripheral neuropathy
* Active or chronic corneal disorder, including but not limited to the following: Sjogren's syndrome, Fuchs corneal dystrophy (requiring treatment), history of corneal transplantation, active herpetic keratitis, and also active ocular conditions requiring on-going treatment/monitoring such as wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, presence of papilledema, and acquired monocular vision
* Serious concurrent illness or clinically-relevant active infection, including, but not limited to the following:

  * Known active hepatitis B or C
  * Known human immunodeficiency virus (HIV) infection
  * Varicella-zoster virus (shingles)
  * Cytomegalovirus infection
  * Any other known concurrent infectious disease, requiring IV antibiotics within 2 weeks of study enrollment
* Clinically-significant cardiac disease:

  * Recent myocardial infarction (=< 6 months prior to day 1)
  * Unstable angina pectoris
  * Uncontrolled congestive heart failure (New York Heart Association > class II)
  * Uncontrolled hypertension (>= Common Terminology Criteria for Adverse Events [CTCAE] version [v]4.03 grade 3)
  * Prior history of hypertensive crisis or hypertensive encephalopathy
  * Uncontrolled cardiac arrhythmias
  * Clinically-significant vascular disease (e.g. aortic aneurysm, or dissecting aneurysm)
  * Severe aortic stenosis
  * Clinically significant peripheral vascular disease
  * >= Grade 3 cardiac toxicity following prior chemotherapy
  * Corrected QT interval (QTc) > 470 for females and > 450 for males
* History of neurological conditions that would confound assessment of treatment-emergent neuropathy
* History of hemorrhagic or ischemic stroke within the last 6 months
* History of cirrhotic liver disease
* Previous clinical diagnosis of non-infectious pneumonitis or non-infectious interstitial lung disease
* Prior hypersensitivity to monoclonal antibodies
* Patients who have a history of another primary malignancy, with the exceptions of: non-melanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for >= 3 years
* Carcinomatous meningitis, untreated central nervous system (CNS) disease or symptomatic CNS metastasis. Patients with previously treated CNS metastasis (excluding carcinomatous meningitis) may participate if they are stable (without evidence of progression by imaging, using identical imaging modality at each assessment, for at least 4 weeks prior to first dose of study treatment), have no evidence of new or emerging CNS metastasis, and are not using steroids for at least 7 days prior to first dose of study treatment
* History or evidence of thrombotic or hemorrhagic disorders within 6 months before first study treatment
* Required used of folate-containing supplements (e.g. folate deficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy L Moulder, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 96 participants signed consent, 54 enrolled during prescreening and 42 enrolled during enrollment, 94 were ineligible due to 4 died prior to starting treatment, 1 found not to be Triple negative breast cancer, 4 withdrew, 73 FR alpha negative, 11 insufficient tissue for analysis of FR alpha and 1 trial closed prior to enrollment.
Groups:
- Cohort A: Advanced Triple-Negative Breast Cancer (TNBC): 6 mg/kg IMGN853 IV Q3W
- Cohort B: Localized Breast Cancer: 6 mg/kg IMGN853 IV Q3W for 4 cycles
Period: Overall Study
Arm/Group | Cohort A: Advanced Triple-Negative Breast Cancer (TNBC) | Cohort B: Localized Breast Cancer
Started | 96 | 0
Completed | 2 | 0
Not Completed | 94 | 0
Not completed — Screen Failure | 94 | 0

BASELINE CHARACTERISTICS:
Population: data provided for 2 participants completed the study for Cohort A; no participants moved to Cohort B
Groups:
- Cohort A: Advanced Triple-Negative Breast Cancer(TNBC): 6 mg/kg IMGN853 IV Q3W
Arm/Group | Cohort A: Advanced Triple-Negative Breast Cancer(TNBC)
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 40 [39 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Metastatic Participants With Radiographic Response
Description: Determine if Mirvetuximab Soravtansine as a Single Agent is Likely to Induce Response in at Least 20% of Patients With Metastatic Folate Receptor (FR) Alpha+ Triple Negative Breast Cancer (TNBC). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From the registration to the study until disease progression or death from any cause, whichever occurred first, assessed up to 2 years
Population: We did not enroll enough patients to determine if 20% of patients with metastatic FR+ had a response to mirvetuximab soravtansine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Advanced Triple-Negative Breast Cancer (TNBC)
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Number of Neoadjuvant Participants With Pathologic Response
Description: Determine if mirvetuximab soravtansine as a single agent in the neoadjuvant setting will improve rates of excellent pathologic response (pathologic complete response [pCR]/residual cancer burden [RCB]-0 or RCB-I) from 5% to 20% in patients with high risk, chemotherapy insensitive, FRalpha+ TNBC.
Time Frame: From baseline to the study until disease progression or surgery, assessed up to 6 months
Population: We did not enroll patients in this cohort and no data was collected for this cohort.
Arm/Group | Cohort B: Localized Breast Cancer
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Radiographic Response Rate
Description: Tumor response for patients with measurable lesions should be assessed using RECIST 1.1 (Eisenhauer 2009, 0). Patients with measurable lesions should be assessed using CT or MRI scan approximately every second cycle, from the date of first dose until the 30-day Follow-up visit. Although progression may be determined by the investigator based upon clinical deterioration, every effort should be made to document progression using radiographic methods. The basis for determination of progression per clinical deterioration should be documented.
Time Frame: From the baseline to the study until disease progression or death from any cause, whichever occurred first
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Advanced Triple-Negative Breast Cancer (TNBC)
Number analyzed (Participants) | 2
Participants | 2

4. Secondary Outcome: Number of Participants With Stable Disease
Time Frame: From the baseline to the study until disease progression or death from any cause, whichever occurred first
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Advanced Triple-Negative Breast Cancer (TNBC)
Number analyzed (Participants) | 2
Participants | 1

5. Secondary Outcome: Number of Participants With Progressive Disease
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the baseline to the study until disease progression or death from any cause, whichever occurred first
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Advanced Triple-Negative Breast Cancer (TNBC)
Number analyzed (Participants) | 2
Participants | 1

6. Secondary Outcome: Number of Metastatic Participants With Duration of Response
Description: Determine duration of response metastatic TNBC patients treated with mirvetuximab soravtansine .
Time Frame: From the date of enrollment/baseline of the study until disease progression or death from any cause, whichever occurred first, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Advanced Triple-Negative Breast Cancer (TNBC)
Number analyzed (Participants) | 2
Participants | 2

7. Secondary Outcome: Compare Participants Disease Response FRalpha+ Chemotherapy Resistant Disease vs Similar Molecular Features Who Receive Standard Taxane-based Chemotherapy
Description: Compare disease response (as measured by pCR/RCB-I) in patients with FRalpha+ chemotherapy resistant disease treated on clinical trial with mirvetuximab soravtansine in the neoadjuvant setting to those with similar molecular features who receive standard taxane-based chemotherapy as the second phase of their NACT
Time Frame: From the date of enrollment/baseline of the study until disease progression or death from any cause, whichever occurred first
Population: We did not enroll patients in cohort A and no data was collected for this cohort.
Arm/Group | Cohort A: Advanced Triple-Negative Breast Cancer (TNBC)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected from the initiation of study drugs up to last dose of study drugs, up to 2 years
Arm/Group | Cohort A: Advanced Triple-Negative Breast Cancer (TNBC)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Advanced Triple-Negative Breast Cancer (TNBC) (N=2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Grade 1 Blurred Vision (Eye disorders) | 1 (1)
Grade 2 Blurred Vision (Eye disorders) | 1 (1)
Keratopathy (Eye disorders) | 1 (1)
Peripheral (Nervous system disorders) | 1 (1)
Neutropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03106077/Prot_SAP_001.pdf